CLINICAL TRIAL: NCT05495269
Title: Pilot, Open-label Study of Safety and Tolerability of QLS-101 in Adolescents With Sturge-Weber Syndrome (SWS)-Related Glaucoma Due to Elevated Episcleral Venous Pressure (EVP)
Brief Title: Safety and Tolerability Study of QLS-101 in Adolescents With Sturge-Weber Syndrome (SWS)-Related Glaucoma Due to Elevated Episcleral Venous Pressure (EVP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qlaris Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QC-205
Record Dates: First submitted 2022-08-02; First posted 2022-08-10 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Sturge-Weber Syndrome; Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Sturge-Weber Syndrome; Glaucoma; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Open-label, single treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- QLS-101, 2.0% (Experimental): Qlaris' investigational product, QLS-101, 2.0% concentration, ocular administration (eye drop), given once daily in the morning to both eyes
  Interventions: Drug: QLS-101 ophthalmic solution, 2.0 %

INTERVENTIONS:
Drug: QLS-101 ophthalmic solution, 2.0 % — ophthalmic solution in a single use dropper vial
  Other Names: QLS-101

SUMMARY:
Open-label study of an investigational product (IP), QLS-101, with 28-day every morning (QAM) dosing to both eyes (OU) in adolescents with SWS who have clinical evidence of glaucoma and/or ocular hypertension (OHT) related to SWS elevated EVP in at least one eye.

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 19 years of age at Screening.
* Diagnosed with SWS
* Elevated IOP
* Willing to continue current dosing regimen of IOP-lowering medications
* Able to provide informed consent and follow study instructions

Exclusion Criteria:

* Expected to undergo IOP-lowering surgery
* Incisional or laser surgery of any type 4 months prior to study
* Ocular infection, inflammation, clinically significant blepharitis or conjunctivitis, history of herpes simplex keratitis in either eye
* History of or active clinically significant ocular disease
* Use of topical ocular corticosteroids in the 6 weeks prior to study
* Patient cannot be applanated or tolerate IOP measurements
* Patient is pregnant or lactating
* Uncontrolled systemic disease that can interfere with study participation
* Inability to self-dose or identify a caregiver for all study eye drop administration

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Ocular safety | Over 28 days
  Incidence of ocular treatment emergent adverse events (TEAEs)
Systemic safety | Over 28 days
  Incidence of systemic TEAEs

SECONDARY OUTCOMES:
Ocular hypotensive effectiveness | 28 days
  Mean change in intraocular pressure (IOP) (mmHg and % change) from baseline following 28 days dosing with QLS-101

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Freedman, M.D., Principal Investigator — Duke Eye Center
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No